CLINICAL TRIAL: NCT07271953
Title: The Effect of Motivational Interviewing and Digital Game-Supported Counseling on Postpartum Relapse in Pregnant Women Who Quit Smoking: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing and Digital Game-Supported Counseling on Postpartum Relapse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Nurbanu Odacı, Lecturer / PhD Candidate in Public Health Nursing, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LokmanHekimU-Hem-NO-02
Record Dates: First submitted 2025-11-23; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Period; Smoking Relapse Behavior
Keywords: Motivational Interviewing; Digital Game; Antenatal care; Smoking relapse
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study with pre-test post-test parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive counseling supported by motivational interviewing and a digital game.
  Interventions: Behavioral: Motivational Interviewing and Digital Game-Supported Counseling
- Control Group (Active Comparator): Participants receive routine antenatal care
  Interventions: Behavioral: Routine Antenatal Care

INTERVENTIONS:
Behavioral: Motivational Interviewing and Digital Game-Supported Counseling — Collaborative, autonomy-supportive counseling delivered in two structured sessions using motivational interviewing techniques, scheduled during the 3rd and 4th routine antenatal visits. The counseling focuses on sustaining abstinence, coping with cues, relapse prevention, and managing partner/household exposure. Each session follows a manualized protocol, with a session checklist completed at every visit. After each session, participants are assigned a digital game-based task designed to reinforce key counseling themes and support behavior maintenance.
  Arms: Intervention Group
Behavioral: Routine Antenatal Care — Routine antenatal care is provided at the study hospital according to the Ministry of Health's pregnancy follow-up program, which includes visits at ≤14 weeks, 18-24 weeks, 28-32 weeks, and 36-38 weeks of gestation.
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to determine the effect of motivational interviewing-based, digital game-supported counseling on postpartum smoking relapse among pregnant women who quit smoking spontaneously during pregnancy. Women who smoked at least one cigarette per day before pregnancy and quit smoking during pregnancy will be included. Participants will be randomly assigned to two groups: in the intervention group, online motivational interviewing sessions will be delivered once each during the third and fourth prenatal follow-ups by the researcher, and a digital game assignment will be provided after each session; the control group will receive routine health counseling delivered during prenatal follow-ups. The primary outcome measure is the rate of smoking relapse at three months postpartum. Secondary outcome measures include the postpartum slip rate, craving to smoke, and motivation to remain abstinent.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Being in the second trimester of pregnancy
* Smoked at least one cigarette per day before pregnancy and quit smoking during the first trimester of pregnancy
* Have internet access
* Own a device capable of playing the digital game (e.g., smart phone, tablet, or computer)
* Native Turkish speakers

Exclusion Criteria:

* Having a diagnosis of any psychiatric disorder
* Currently using another pharmacological or behavioral smoking cessation method
* Having a high-risk pregnancy

Withdrawal Criteria:

* Experience pregnancy termination for any reason
* Do not participate in any stage of the counseling sessions
* Are diagnosed with postpartum depression during the postpartum period
* Resume smoking during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
Point prevalence abstinence | At 3 months postpartum
  7-day point prevalence abstinence at 3 months postpartum
Continuous abstinence | At 3 months postpartum
  Continuous abstinence rate at 3 months postpartum

SECONDARY OUTCOMES:
Motivation for smoking abstinence | At baseline, and at 1, 2, and 3 months postpartum
  Assessed using the Turkish version of the Abstinence-Related Motivational Engagement (ARME) Scale, which evaluates participants' motivation to maintain smoking abstinence through total scale scores.
Level of cigarette craving | At baseline, and at 1, 2, and 3 months postpartum
  Measured using a self-reported 0-10 rating scale for cigarette craving (0 = no craving, 10 = extreme craving).
Prevalence of slips | At 1, 2, and 3 months postpartum
  Prevalence of slips

CONTACTS AND LOCATIONS:
Overall Officials: Bilge KALANLAR, Study Director — Hacettepe Üniversitesi
Locations (1):
- Lokman Hekim Universty, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No